CLINICAL TRIAL: NCT00589251
Title: Equivalency of Penicilloate Skin Test Reactivity Prepared by a Modified Alkaline Hydrolysis Technique
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Miguel Park, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 301-06
Record Dates: First submitted 2007-12-28; First posted 2008-01-09 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Penicillin Allergy
Keywords: penicillin allergy, penicillin skin test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- penicillin skin test (Other): Patients will have the skin test placed
  Interventions: Other: penicillin skin test

INTERVENTIONS:
Other: penicillin skin test — Prick skin tests will be performed on the volar surface of the forearm with each penicilloate and control reagents. The skin test sites will be examined at 15 minutes. A positive test result is defined as a wheal of 3x3 mm or greater with a surrounding zone of erythema. Patients with negative prick test results to penicillin will undergo intradermal testing.
  Intradermal skin tests will be performed on the volar surface of the forearm. The test reagents will be injected intradermally to produce an initial wheal of 2x2 mm. The skin test sites will be examined at 15 minutes. A positive intradermal test is defined as a wheal of 3x3 mm or greater with a surrounding zone of erythema. In order to ensure patient safety, we will consider using an end point titration technique.

SUMMARY:
The primary objective of the study is to evaluate the equivalency of the skin test reactivity to penicilloate prepared by our new method of penicilloate preparation versus our old method of penicilloate preparation. The secondary objective of the study is to evaluate the significance of the different diastereoisomers of penicilloate on skin test reactivity.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the equivalency of the skin test reactivity to penicilloate prepared by our new method of penicilloate preparation versus our old method of penicilloate preparation. The secondary objective of the study is to evaluate the significance of the different diastereoisomers of penicilloate on skin test reactivity.

Five (5) adult subjects without a history of penicillin allergy and fifteen (15) adult subjects with a history of penicillin allergy and previous positive penicillin skin test to the minor determinant (penicilloate) and/or major determinant (penicilloyl) will be enrolled into the study. Each subject will be skin tested with our current penicillin skin test which includes penicilloate conducted in the Division of Allergic Diseases will be compared the skin test of our penicilloate prepared by our newer method along with the different diastereoisomers of penicilloic acid on the same day and time. The adult subjects without a history of penicillin allergy will serve as our control.

ELIGIBILITY:
Inclusion Criteria:

1. History of penicillin allergy
2. Previous or current positive skin test to penicilloate
3. Greater than or equal to 18 years of age

Exclusion Criteria:

1. Uncontrolled asthma by symptoms
2. Patients who have received penicillin and had no adverse drug reaction
3. Previous adverse reaction to penicillin skin test
4. Dermatological conditions that may interfere with skin testing i.e. atopic dermatitis and dermatographism
5. Medication that may interfere with skin testing i.e. antidepressants, antihistamines, and sedatives.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the equivalency of the skin test reactivity to penicilloate prepared by our new method of penicilloate preparation versus our old method of penicilloate preparation. | immediate

SECONDARY OUTCOMES:
The secondary objective of the study is to evaluate the significance of the different diastereoisomers of penicilloate on skin test reactivity. | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Park, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: Undecided